CLINICAL TRIAL: NCT00690131
Title: An Integrated Approach to Smoking Cessation in SMI
Brief Title: An Integrated Approach to Smoking Cessation in Severe Mental Illness (SMI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Melanie Bennett, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00043121; 1R34MH080814-01A1 (NIH)
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Smoking Cessation
Keywords: Smoking cessation, severe mental illness, behavioral treatment
MeSH Terms: conditions — Smoking Cessation; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: BTSCS
- 2 (No Intervention)

INTERVENTIONS:
Behavioral: BTSCS — BTSCS includes: (1) A behavioral group emphasizing motivational enhancement, skills training, education, and relapse prevention; (2) Contingency management with financial incentives to reinforce reductions in smoking; (3) Supported use of Bupropion or nicotine replacement therapy that is integrated with clients' psychiatric care in participants who are interested; and (4) Smoking cessation care coordination to increase treatment engagement and retention.
  Arms: 1

SUMMARY:
This 3-year study will involve the design and small-scale clinical trial of a behavioral treatment program for smoking cessation in people with severe mental illness (called Behavioral Treatment for Smoking Cessation in Serious and Persistent Mental Illness or BTSCS) in two psychosocial rehabilitation programs (PRPs) in Baltimore. Our aims are: (1) Develop intervention materials and examine feasibility, acceptability, and safety; (2) Measure the effects of the intervention at post-treatment and 3-month follow-up on rates of smoking cessation, number of quit attempts, rates of smoking reduction and intention/motivation to quit smoking.

DETAILED DESCRIPTION:
Smoking is the leading cause of preventable death in the United States, contributing to increased rates of lung cancer and heart disease, and adding complications to other health problems. Over 70% of people with serious mental illnesses (SMI) smoke, a rate that is double that of the general population and remains high despite decreases in overall smoking rates. Smoking contributes to elevated morbidity and mortality in SMI, has other life-threatening consequences, and increases health care costs in SMI. While treating smoking is a critical step in improving the health of people with SMI, there are features of SMI that make treatment difficult (low motivation to quit, symptoms, barriers to attendance, cognitive deficits, poor social functioning). Stop-smoking groups have had limited success in achieving smoking cessation (SC), likely because they have not been tailored for people with SMI. SC for SMI must address the deficits and barriers to change found in this population, and must be integrated with mental health services.

This study will involve the design and small-scale clinical trial of a behavioral treatment program for SC in people with SMI called Behavioral Treatment for Smoking Cessation in Serious and Persistent Mental Illness (BTSCS) in two psychosocial rehabilitation programs (PRPs) in Baltimore.

We will first provide basic education for PRP staff regarding smoking cessation in SMI to promote smoking cessation as a goal of mental health treatment. We will then pilot test BTSCS with components that include: (1) A behavioral group emphasizing motivational enhancement, skills training, education, and relapse prevention; (2) Contingency management with financial incentives to reinforce reductions in smoking; (3) Supported use of Bupropion or nicotine replacement therapy that is integrated with clients' psychiatric care in participants who are interested; and (4) Smoking cessation care coordination to increase treatment engagement and retention. Our primary aims are: (1) Develop intervention materials and examine feasibility, acceptability, and safety; (2) Measure the effects of the intervention at post-treatment and 3-month follow-up on rates of smoking cessation, number of quit attempts, rates of smoking reduction and intention/motivation to quit smoking.

ELIGIBILITY:
Inclusion Criteria:

* Severe and Persistent Mental Illness (schizophrenia, schizoaffective disorder or other severe mental disorder including bipolar disorder, major depression, or severe anxiety disorder).
* Age between 18 and 75 years.
* Current smokers who smoke at least 10 cigarettes per day.
* Must have been seen by a psychiatrist at least every 3 months for the last 6 months.

Exclusion Criteria:

* Meet criteria for current alcohol/substance dependence (other than nicotine).
* Documented mental retardation, history of severe head injury with LOC, severe and untreated seizure disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Smoking abstinence: percentage of participants reporting abstinence reported in the 7-day interval at post-treatment and follow-up | 7-day interval at post-treatment and follow-up
Smoking abstinence: average percentage of biweekly sessions with negative expired carbon monoxide (CO) levels (< 8 ppm) | from baseline to post treatment
Number of smoking quit attempts: self-reported number of quit attempts (for at least 24 hours) at post treatment and 3 month follow-up | time from baseline to post treatment and baseline to 3 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Melanie E Bennett, Ph.D., Principal Investigator — University of Maryland, College Park
Locations (3):
- United States (3):
  - University of Maryland Baltimore, Baltimore, Maryland
  - Harbor City Unlimited, Baltimore, Maryland
  - New Ventures, Sheppard Pratt, Timonium, Maryland